CLINICAL TRIAL: NCT05388929
Title: Addition of Methocarbamol to Postoperative Multimodal Analgesic Regimen: A Prospective, Randomized Pilot Study
Brief Title: Methocarbamol in Ventral and Inguinal HR
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1913843
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Ventral Hernia; Inguinal Hernia
MeSH Terms: conditions — Hernia, Ventral; Hernia, Inguinal | interventions — Methocarbamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- primary ventral hernia repair or inguinal hernia repair (Experimental): Primary ventral hernias, including umbilical, epigastric, and Spigelian hernias.
  Primary or recurrent inguinal hernias.
  Interventions: Drug: Methocarbamol; Drug: Standard Opioid
- open or robotic ventral hernia repair outpatient (Experimental): Open repair of ventral incisional hernias. Robotic repair of ventral primary or incisional hernias.
  Interventions: Drug: Standard Opioid; Drug: Standard opioid plus methocarbamol
- open or robotic hernia repair inpatient (Experimental): Open repair of ventral incisional hernias. Robotic repair of ventral primary or incisional hernias.
  Interventions: Drug: Standard Opioid; Drug: Standard opioid plus methocarbamol

INTERVENTIONS:
Drug: Methocarbamol — Methocarbamol after surgery
  Arms: primary ventral hernia repair or inguinal hernia repair
Drug: Standard Opioid — Standard opioid after surgery or at discharge
Drug: Standard opioid plus methocarbamol — Standard opioid plus methocarbamol after surgery or at discharge
  Arms: open or robotic hernia repair inpatient; open or robotic ventral hernia repair outpatient

SUMMARY:
The purpose of this study is to gather information on methocarbamol as a pain management treatment for ventral or inguinal hernia repair.

Methocarbamol has been part of the pain management treatment for both inpatient and outpatient procedures at Prisma Health. This study will compare the outcomes of patients who receive methocarbamol, those who receive the standard opioid pain management treatment, and those who receive methocarbamol plus the standard opioid pain management treatment.

Participants will be randomized into one of the study groups listed below.

Primary ventral hernia repair or inguinal hernia repair:

Group 1: standard opioid after surgery Group 2: methocarbamol after surgery

Open or robotic ventral hernia repair outpatient:

Group 1: standard opioid after surgery Group 2: standard opioid plus methocarbamol after surgery

Open or robotic ventral hernia repair inpatient:

Group 1: standard opioid at discharge Group 2: standard opioid plus methocarbamol at discharge

A total of 200 participants will be included in the study.

Participation will last for about 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* >18 y/o
* Patients undergoing open primary ventral hernia repair (group 1)
* Patients undergoing inguinal hernia repair (open, laparoscopic, or robotic; group 2)
* Patients undergoing open incisional hernia repair (group 3)
* Robotic repair ventral or incisional hernias (group 4)
* Given consent for randomization

Exclusion Criteria:

* <18 y/o
* Pregnancy
* Chronic opioid users

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients requiring a rescue opioid prescription | 30 days post surgery
  The proportion of patients requiring a rescue opioid prescription will be compared between the study and control groups using the Fisher's Exact Test (bivariate analysis). Multiple logistic regression analysis will then be used to test for a difference in this outcome, adjusting for any baseline differences between the 2 study groups.
Average total morphine milligram equivalents (MME) consumption | 30 days post surgery
  Average total MME consumption will be compared between the study and control groups using either the Student's T-test or the Wilcoxon Rank Sum Test (depends on distribution of the data -- parametric vs. non-parametric).

SECONDARY OUTCOMES:
European Registry of Abdominal Wall Hernias (EuraHS) Quality of Life tool scores | 30 days post surgery
  Scale of 0-10, where 0 = no pain and 10 = worst pain imaginable. Outcome will be compared between the study and control groups using either the Student's T-test or the Wilcoxon Rank Sum Test. Statistical tests used are dependent on the data distribution -- parametric vs. non-parametric).
Visual Analog Scale pain scores | 7 days post surgery
  Scale of 0-10, where 0 = no pain and 10 = worst pain imaginable. Outcome will be compared between the study and control groups using either the Student's T-test or the Wilcoxon Rank Sum Test. Statistical tests used are dependent on the data distribution -- parametric vs. non-parametric).

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy A Warren, MD, Principal Investigator — Prisma Health
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No